CLINICAL TRIAL: NCT04974502
Title: The Influence of Smoking on Oral Neutrophils and Matrix Metalloproteinase-8 in Periodontitis Patients, Before and After Nonsurgical Treatment
Brief Title: The Influence of Smoking in Periodontitis Patients, Before and After Nonsurgical Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Nguyen Thu Thuy, Associate Dean of Faculty of Odonto-stomatology, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 92/DHYD-HDDD
Record Dates: First submitted 2021-07-01; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Periodontitis
Keywords: periodontitis; smoking; neutrophil; matrix metalloproteinase-8; nonsurgical treatment
MeSH Terms: conditions — Periodontitis; Smoking

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-smoker group (Experimental)
  Interventions: Procedure: Nonsurgical periodontal treatment
- Smoker group (Experimental)
  Interventions: Procedure: Nonsurgical periodontal treatment

INTERVENTIONS:
Procedure: Nonsurgical periodontal treatment — Oral hygiene instructions, scaling and root planning.

SUMMARY:
Objective: The aim of this study was to evaluate and compare the oral neutrophil numbers (ONN) in saliva, the level of matrix metalloproteinase-8 (MMP-8) in gingival crevicular fluid (GCF) and the periodontal parameters in smokers and non-smokers with periodontitis, before and after nonsurgical periodontal treatment (NSPT).

Materials and method: 40 periodontitis patients including 20 smokers and 20 non-smokers were enrolled in this study. All patients were received the NSPT included instructing oral hygiene, scaling and root planning. Clinical parameters (plaque index (PlI), gingival index (GI), bleeding on probing (BOP), probing pocket depth (PPD) and clinical attachment loss (CAL)), ONN and GCF MMP-8 level were assessed before (baseline) and after NSPT 1 month and 3 months.

DETAILED DESCRIPTION:
After periodontal examination and medical history evaluation, all patients received oral hygiene instructions. The modified-Bass tooth brushing technique, as well as the use of dental floss and interproximal brushes (if needed) were showed to the patients. They were educated to brush their teeth at least twice a day. All patients were given a dentifrice and toothbrush. Patient motivation to quit smoking was also provided.

At the first visit, supragingival scaling with ultrasonic scalers (Cavitron Jet Plus (Densply Sirona, Mississauga, Canada) were provided to all patients. Occlusion adjustments were also performed in the case of indications.

After one week, the baseline (T0) parameters were recorded. The following samples were collected: (1) saliva, (2) gingival cervical fluid (GCF), and (3) clinical periodontal parameters. A doctor who collected the samples was blinded about the smoking status.

Subsequently, scaling and root planning (SRP) by ultrasonic scalers (Cavitron Jet Plus (Densply Sirona, Mississauga, Canada) and Gracey curettes (Hu-Friedy, Chicago, USA), under local anesthesia, were performed by a periodontist, who was also blinded about the smoking status. The number of SRP visits was determined by patient disease conditions.

Following the completion of NSPT, all subjects were recalled after one month and three months for re-evaluation. The collection of (1) saliva, (2) gingival cervical fluid (GCF), and (3) clinical periodontal parameters were performed. Based on the patients' periodontal status, supragingival scaling and polishing were given.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Aged from 30 to 60 years old
* Systemically healthy
* Having at least 20 teeth
* Diagnosed with moderate to severe periodontitis according to american academy of periodontology 2015: gingival bleeding at examination, ≥5mm periodontal pocket depth (PPD), bone resorption on x-ray film ≥16% or >3mm root length
* Having at least two sites at anterior teeth with PPD from 5 to 7 mm
* For group 1, subjects who never smoke
* For group 2, subjects who had smoked more than 10 cigarettes per day for at least the past 10 years

Exclusion Criteria:

* Patients with acute or chronic medical disorders
* Patients under any medication for the past 3 months
* Patients who had undergone periodontal therapy in the last 12 months
* Patients with oral lesions such as ulcers, aphthous ulcers, glossitis or multi tooth decays

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Smoking male
Enrollment: 40 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Oral neutrophils | At baseline (T0)
  The number of neutrophils in saliva
Oral neutrophils | After Nonsurgical periodontal treatment one month (T1)
  The number of neutrophils in saliva
Oral neutrophils | After Nonsurgical periodontal treatment three months (T3)
  The number of neutrophils in saliva
Matrix metalloproteinase-8 (MMP-8) | At baseline (T0).
  The level of matrix metalloproteinase-8 (MMP-8) in gingival crevicular fluid
Matrix metalloproteinase-8 (MMP-8) | After Nonsurgical periodontal treatment three months (T3)
  The level of matrix metalloproteinase-8 (MMP-8) in gingival crevicular fluid

SECONDARY OUTCOMES:
Plaque Index (PlI) | At baseline (T0).
  Plaque Index (Silness and Loe, 1967)
Plaque Index (PlI) | After Nonsurgical periodontal treatment one month (T1)
  Plaque Index (Silness and Loe, 1967)
Plaque Index (PlI) | After Nonsurgical periodontal treatment three months (T3)
  Plaque Index (Silness and Loe, 1967)
Gingival Index (GI) | At baseline (T0).
  Gingival Index (Silness and Loe, 1967)
Gingival Index (GI) | After Nonsurgical periodontal treatment one month (T1)
  Gingival Index (Silness and Loe, 1967)
Gingival Index (GI) | After Nonsurgical periodontal treatment three months (T3)
  Gingival Index (Silness and Loe, 1967)
Probing pocket depth (PPD) | At baseline (T0).
  The distance from the gingival margin to pocket base
Probing pocket depth (PPD) | After Nonsurgical periodontal treatment one month (T1)
  The distance from the gingival margin to pocket base
Probing pocket depth (PPD) | After Nonsurgical periodontal treatment three months (T3)
  The distance from the gingival margin to pocket base
Clinical attachment loss (CAL) | At baseline (T0).
  The distance from the cementoenamel junction (CEJ) to the gingival margin
Clinical attachment loss (CAL) | After Nonsurgical periodontal treatment three months (T3)
  The distance from the cementoenamel junction (CEJ) to the gingival margin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al-Ghamdi HS, Anil S. Serum antibody levels in smoker and non-smoker saudi subjects with chronic periodontitis. J Periodontol. 2007 Jun;78(6):1043-50. doi: 10.1902/jop.2007.060431. PMID 17539718
- [Result] Akbari G, Prabhuji ML, Karthikeyan BV, Raghunatha K, Narayanan R. Analysis of matrix metalloproteinase-8 levels in gingival crevicular fluid and whole mouth fluid among smokers and nonsmokers using enzyme-linked immune-sorbent assay and a novel chair-side test. J Indian Soc Periodontol. 2015 Sep-Oct;19(5):525-30. doi: 10.4103/0972-124X.162201. PMID 26644719
- [Derived] Do HT, Nguyen TT, Vo TL, Huynh NC, Nguyen ATK. The influence of smoking on oral neutrophils and matrix metalloproteinase-8 in periodontitis patients before and after nonsurgical treatment. J Oral Biol Craniofac Res. 2023 May-Jun;13(3):442-447. doi: 10.1016/j.jobcr.2023.05.004. Epub 2023 May 8. PMID 37215391